CLINICAL TRIAL: NCT06440473
Title: Visualization of Topical Zoryve vs. Vehicle Using Line Field Optical Coherence Tomography in Healthy Skin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rao Dermatology (Other)
Responsible Party: Principal Investigator, Babar Rao, Principal Investigator and Owner, Rao Dermatology
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00078950
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Skin
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast (Active Comparator)
  Interventions: Drug: Roflumilast
- Vehicle (Placebo Comparator)
  Interventions: Other: Vehicle (Roflumilast 0.3% vehicle cream)

INTERVENTIONS:
Drug: Roflumilast — Roflumilast 0.3% cream
  Arms: Roflumilast
Other: Vehicle (Roflumilast 0.3% vehicle cream) — Vehicle (Roflumilast 0.3% vehicle cream)
  Arms: Vehicle

SUMMARY:
The goal of this study is to visualize the deposition of topical 0.3% roflumilast (Zoryve) compared to vehicle using Line-Field Optical Coherence Tomography (LC-OCT) in vivo in healthy skin. We hypothesize that the application of topical 0.3% roflumilast (Zoryve) will result in distinct patterns of deposition within the epidermal and dermal layers compared to the vehicle. Specifically, we anticipate observing deeper penetration and more uniform distribution of roflumilast within the skin layers, indicative of enhanced efficacy, as visualized by LC-OCT imaging.

DETAILED DESCRIPTION:
Primary Objective

Compare the deposition of Zoryve and the vehicle in the epidermal and dermal layers using LC-OCT.

Primary Endpoint

The primary endpoint of this study is a visual qualitative analysis of LC-OCT images conducted by an expert confocalist, Babar Rao MD. This analysis aims to assess the penetration of the active drug product compared to the vehicle.

Subjects will be instructed to apply topical 0.3% Zoryve once daily for seven consecutive days to a predetermined 2x2cm area on the dorsal surface forearm, as defined by the investigator. Additionally, participants will apply a topical cream vehicle provided by Zoryve to the dorsall side of the opposite forearm. Therefore, one forearm, will be designated for application of Zoryve, while the other forearm will the designated for application of the topical cream vehicle supplied by Zoryve. Subjects will apply the topical vehicle and roflumilast, daily, for 7 consecutive days. LC-OCT imaging will be conducted on both arms at various time points: baseline (T0A), 15 minutes (T0B), 1 hour (T0C), 8-12 hours (T0D), 24 hours (T0E), seven days after application (T7), and seven days after not applying cream (T14). LC-OCT imaging will follow a predefined image acquisition protocol, with investigators designating 2x2cm areas for imaging. The imaging protocol will include capturing 2D vertical photos, 3D photos, and 2D vertical videos per imaging site. Participants will be instructed to photograph the imaging sites to aid in the accurate application of the active drug product or vehicle cream base.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 18 years of age from the outpatient dermatology clinic, Rao Dermatology. All subjects must have provided written informed consent.

Exclusion Criteria:

* Subjects with a history of immune-mediated skin conditions will be excluded from participation. Additionally, participants who have received systemic therapy within the last 60 days will not be eligible. Those using topical therapy must have discontinued their current treatment for a minimum of seven days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-05-28 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
LC-OCT | 14 days
  The primary endpoint of this study is a visual qualitative analysis of LC-OCT images conducted by an expert confocalist, Babar Rao MD. This analysis aims to assess the penetration of the active drug product compared to the vehicle.

CONTACTS AND LOCATIONS:
Locations (1):
- Rao Dermatology, Atlantic Highlands, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Results to be reported as pulled data

REFERENCES:
- [Background] Pixley JN, Schaetzle T, Feldman SR. A Review of Topical Roflumilast for the Treatment of Plaque Psoriasis. Ann Pharmacother. 2023 Aug;57(8):966-969. doi: 10.1177/10600280221137750. Epub 2022 Nov 24. PMID 36420929